CLINICAL TRIAL: NCT06769022
Title: Exercise Adherence and Cognitive Decline: Engaging With the Black Community to Develop and Test a Goal-Setting and Exercise Intensity Intervention
Brief Title: Exercise Adherence and Cognitive Decline
Acronym: MOVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Angela Bryan, PI, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-01-0205; 1R61AG078088-01A1 (NIH)
Record Dates: First submitted 2024-12-03; First posted 2025-01-10 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Decline
Keywords: Goals; Exercise Intensity; Goal Difficulty; Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Moderate Intensity Exercise, Basic Goal Difficulty (Experimental): Participants are assigned to exercise at a moderate intensity and create basic goals.
  Interventions: Behavioral: Goal Setting and Exercise Intensity Intervention
- Moderate Intensity Exercise, Challenging Goal Difficulty (Experimental): Participants are assigned to exercise at a moderate intensity and create challenging goals.
  Interventions: Behavioral: Goal Setting and Exercise Intensity Intervention
- Vigorous Intensity Exercise, Basic Goal Difficulty (Experimental): Participants are assigned to exercise at a vigorous intensity and create basic goals.
  Interventions: Behavioral: Goal Setting and Exercise Intensity Intervention
- Vigorous Intensity Exercise, Challenging Goal Difficulty (Experimental): Participants are assigned to exercise at a vigorous intensity and create challenging goals.
  Interventions: Behavioral: Goal Setting and Exercise Intensity Intervention

INTERVENTIONS:
Behavioral: Goal Setting and Exercise Intensity Intervention — Participants' goal-setting and exercise intensity are manipulated based on group assignment.

SUMMARY:
The purpose of this study is to conduct a small-scale test of a goals-based program to help people to exercise more and learn what people like or don't like about the procedures. This program is being designed for individuals aged 45-65 from the Black community. Low levels of physical activity are related to health problems such as heart disease, diabetes, and cognitive decline. People of color are more negatively impacted by these conditions and have also historically been underrepresented by research seeking to increase physical activity. The investigators have developed this goals-based exercise promotion program with the help of a Black-led community-based organization (The Gyedi Project) and a Community Advisory Board made up of stakeholders in the Black community, and now the investigators are conducting a trial of its feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* <3 incorrect responses on the Pfeiffer Mental Status Questionnaire
* Ages 45-65.
* Consent to be randomized to condition.
* Planning to remain in the Denver metro area for the next two months
* Identify as Black or African American

Exclusion Criteria:

* Currently physically active (i.e., >90 min/week of moderate PA or >40 min/week of vigorous PA consistently for the past 6 months).
* On antipsychotic medications or currently under treatment for any serious psychiatric disorder, including Alzheimer's or dementia
* Answers "yes" to 1 or more of the 7 questions of the PAR-Q+
* Blood pressure at baseline or before exercise is greater than 140/90
* Blood pressure >210/90 mmHg (for men) or >190/90 mmHg (for women) immediately after exercise
* Inability to walk 3 blocks without chest pain, shortness of breath, or light headedness.
* Inability to climb 2 flights of stairs without chest pain, shortness of breath, or light headedness.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Baseline, Visit 14 (~2 months after baseline)
  Blood pressure of all participants is collected before intervention
Activity Levels | Baseline, Visit 14 (~2 months after baseline)
  Exercise Intensity (PAR). Answers are direct (ex. how many hours active) and not scaled. Information is requested for the week and the past 3 months.
Sleep levels | Baseline, Visit 14 (~2 months after baseline)
  Exercise Intensity (PAR). Answers are direct (ex. how many hours did you sleep) and are not scaled. Information is requested for the past 7 days.
Physical Activity Recall | Baseline, Visit 14 (~2 months after baseline)
  Exercise Intensity (PAR). Answers are direct (ex. how many hours did you sleep) and are not scaled. Information is requested for the past 7 days.
Identity | Baseline
  Multidimensional Black Identity Scale to collect information on identity. Questions are about personal identity relating to the Black community on a scale of 1-7, 1 being strongly disagree and 7 being strongly agree. Higher scores indicate a stronger agreement with that dimension of Black identity. Scores are summed as subscales and averaged to obtain an average score.
Exercise Behavior | Baseline, Visit 14 (~2 months after baseline)
  CHAMPS. The survey collects quantitative data looking at the approximate total hours per week spent doing various activities, both physical and social.
Exercise Behavior | Baseline, Visit 14 (~2 months after baseline)
  L-Cat. Single question that asks about frequency/rigor of physical activity, with six potential answers ranging from no physical activity to daily physical activity.
Theoretical Mediators of Exercise Behavior | Baseline, Visit 12 (~1 month after baseline), Visit 14 (~2 months after baseline)
  Intrinsic Motivation Inventory. Questions relate to how participants think or feel about physical activity, with answers ranging from 1 (strongly disagree) to 7 (strongly agree). Broader scores are broken up into subscales; final subscale scores are summed and averaged. Higher scores indicate higher agreement with that subscale.
Theoretical Mediators of Exercise Behavior | Baseline, Visit 12 (~1 month after baseline), Visit 14 (~2 months after baseline)
  Self-Efficacy. 9 questions about confidence in exercise on scale of 1 (disagree strongly) to 7 (agree strongly). Higher scores indicate higher perceived confidence in doing that activity. Total scores are summed.
Theoretical Mediators of Exercise Behavior | Baseline, Visit 12 (~1 month after baseline), Visit 14 (~2 months after baseline)
  Exercise Intention Survey. Scored on a Likert scale from 1 (strongly disagree) to 7 (strongly agree) to indicate level of agreement to statements related to intention to exercise. Scores are summed to produce a total score. Higher scores indicate stronger intention to exercise, lower scores indicate weaker intention.
Theoretical Mediators of Exercise Behavior | Baseline, Visit 12 (~1 month after baseline), Visit 14 (~2 months after baseline)
  Exercise Identity Score. Scored on a Likert scale from 1 (strongly disagree) to 7 (strongly agree) to indicate level of agreement to statements related to attitudes towards exercise. Scores are summed and averaged to provide an overall score. Higher scores indicate a positive attitude towards exercise, lower scores less favorable attitude.
Heart Rate Variability | Baseline, Visit 14 (~2 months after baseline)
  Heart Rate Variability is measured using chest strap monitor.
Heart Rate | Baseline, Visits 1-14 (all visits)
  HR is measured using chest strap monitor.
Physical Performance | Baseline, Visit 14 (~2 months after baseline)
  Short Physical Performance Battery. Physical performance measured with repeated chair stands, three balance tests (side-by-side, semi-tandem, tandem), timed walking.
Ventilatory Threshold | Baseline
  Talk Test. Graded treadmill test where intensity is increased at intervals to determine participant's ventilatory threshold.
Perceived Exertion | Visit 2-13 (~2 visits/week)
  A single-item measure from Borg (1973) was used to assess participants' rate of perceived exertion (RPE) during the exercise bout. Participants were asked to rate the average intensity of exercise [at that moment/during the past ten minutes] on a 25-point scale ranging from 6 (no exertion at all) to 20 (maximal exertion).
Pain Levels | Visit 2-13 (~2 visits/week)
  A single item measure from Borg (1998) was used to assess participants' pain levels during the exercise bout. Participants were asked to indicate how much pain they felt [at that moment/during the past ten minutes] on an 11-point scale ranging from 0 (nothing at all) to 10 (excruciating).
Affective Valence | Visit 2-13 (~2 visits/week)
  The Feeling Scale, a single-item measure from Hardy and Rejeski (1989), was used to assess participants' affective valence during the exercise bout. Participants were asked to indicate how they felt [at that moment/during the past ten minutes] on an 11-point scale ranging from -5 (very bad) to +5 (very good).
Affective Arousal | Visit 2-13 (~2 visits/week)
  The Felt Arousal Scale, a single-item measure from Svebak and Murgatroyd (1985), was used to assess participants' affective arousal during the exercise bout. Participants were asked to indicate how "worked-up" they felt [at that moment/during the past ten minutes] on a 6-point scale ranging from 1 (low arousal) to 6 (high arousal).
Enjoyment | Visit 2-13 (~2 visits/week)
  A single item measure from Gillman and Bryan (2015) was used to assess participants' enjoyment levels during the exercise bout. Participants were asked to indicate how enjoyable exercise was [at that moment/during the past ten minutes] on a 5-point scale ranging from 1 (no enjoyment at all) to 5 (a great deal of enjoyment).
Exercise Check-In | Daily between visit 13 and 14 (~1 month)
  Three short questions assessing if the participant planned to engage in exercise and how many minutes of moderate (0-120) and vigorous (0-60) exercise they engaged in
Study Feedback | Visit 14 (~2 months after baseline)
  An investigator led interview to pilot study participants' experience of the intervention and suggestions for improvement
Exercise Benefits and Barriers | Baseline, Visit 12 (~1 month after baseline), Visit 14 (~2 months after baseline)
  A 10 item scale assessing perceived benefits of and barriers to exercise
Anthropometrics | Baseline
  Height, weight, waist circumference, and hip circumference will be measured
Exercise Aligned with Black Identity | Baseline
  Assessment of the extent to which 7 common exercises are aligned with Black identity
Mental Status | Baseline
  Pfeiffer Mental Status. Assessment of cognitive deficits at baseline.
Diet | Baseline
  Nutrition Data System for Research (NDSR) 24-Hour Dietary Recall. Interviewer administered recall developed by the University of Minnesota Nutrition Coordinating Center (NCC).
Diet | Baseline
  NCI's Eating at America's Table Study (EATS) Fruit & Vegetable All-Day Screener174
  NCI's Eating at America's Table Study (EATS) Fruit & Vegetable All-Day Screener174 NCI's Eating at America's Table Study (EATS) Fruit & Vegetable All-Day Screener. A short dietary assessment instrument for measuring fruit and vegetable intake over the past month.
Physical Activity | Baseline
  Godin Survey. This survey measures time spent in moderate, strenuous or light activity and has been modified to include time spent sitting over a typical 7 day period. Scores are summed and a range is used to quantify how active/sedentary a participant is.

SECONDARY OUTCOMES:
Demographics | Baseline
  Survey includes sex assigned at birth, gender identity, sexual orientation, age, detailed race/ethnicity, and SES

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Aurora Center for Active Adults, Aurora, Colorado
  - University of Colorado at Boulder, Boulder, Colorado
  - Hiawatha Davis Jr. Recreation Center, Denver, Colorado